CLINICAL TRIAL: NCT03883594
Title: Technology Assisted Stepped Care (TASC): Phase 3
Brief Title: Technology-Assisted Stepped Care Study
Acronym: TASC Phase 3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CIN001- {"TASC Phase 3"}
Record Dates: First submitted 2019-02-08; First posted 2019-03-21 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TASC Intervention (Experimental): All participants receive Step 1 of the intervention. Participants who have adherence below or at 68% will step up to Step 2 or Step 3 after the third or fourth month in the study.
  Interventions: Behavioral: Technology-assisted Stepped-care

INTERVENTIONS:
Behavioral: Technology-assisted Stepped-care — Step 1 of the intervention includes educational materials related to asthma. Step 2 includes electronic monitoring of adherence and a text messaging intervention personally tailored to the participant. Step 3 includes problem solving telehealth sessions with a trained clinician.

SUMMARY:
The overall goal of this project is to demonstrate the feasibility, implementation, and preliminary efficacy of a technology-assisted stepped care (TASC) adherence-promotion intervention in adolescents with asthma. This is the third phase (Phase 3) of a three-phase project to test the preliminary efficacy of a technology-assisted stepped care (TASC) intervention. In Phase 1, we developed the intervention using patient and provider feedback from focus groups. In Phase 2 we refined the developed intervention by having five adolescents from the focus groups test the intervention for feasibility. In this third phase, we will enroll up to 50 adolescents to pilot-test the refined intervention for preliminary efficacy.

DETAILED DESCRIPTION:
Up to fifty adolescents with asthma will be enrolled in an open label pilot trial of the TASC adherence-promotion intervention for a duration of twelve months. First, participants will complete baseline questionnaires related to demographic, and clinical predictors of adherence and asthma and a 4 week run-in phase to assess baseline adherence using electronic inhaler monitoring with a cellphone that is provided to them. Following the run-in period, all participants will receive Step 1 of the TASC intervention for a minimum of 4 weeks. Step 1 (Information) will include electronic educational information related to asthma symptoms and triggers, attacks, self-monitoring, treatments, action plans, and automated text message medication reminders. Following the initial four weeks of Step 1, adherence will be evaluated and a rate of less than 68% will serve as the cause for "stepping up" to the next level of the intervention. Adherence checks will continue to occur every four weeks for the duration of the study and adherence <68% will prompt movement from one level of treatment to the next. Participants may remain at a treatment level for more than four weeks and may complete 1, 2, or 3 interventions steps during the 5 month study depending on the adolescent's adherence. Step 2 (Motivation) will include electronic monitoring of adherence and personally tailored feedback via text messages. Adolescents will be given access to the adherence tracking cellphone app and graphs of their inhaler adherence. Adolescents will also receive brief, personalized text messages that provide supportive motivation and directive, tangible actions. Step 3 (Behavioral) will include problem-solving telehealth intervention with a trained clinician. Four telehealth sessions individually tailored to the unique needs and barriers of the adolescent will be provided. The primary outcome measure will be electronically-monitored adherence assessed at post-treatment. Secondary outcomes include asthma severity as well as process evaluation questions and quantitative measures of feasibility, acceptability, and satisfaction to demonstrate implementation. Participants will remain in the study for an additional 7 months after they complete month 5 of the study. For the remaining 7 months, participants will be randomized to one of two booster session patterns with the goal to improve inhaler adherence. The statistician will make the randomization schedule and the principle investigator will maintain the randomization schedule. Two different booster patterns are being used to test which pattern will be most effective. The first booster session pattern will include booster sessions at the end of month 6, 8, and 12. The second booster session pattern will include booster sessions at the end of month 6, 7, 8, 10, and 12. Booster sessions will review content provided during the intervention and the intervention delivery method will be consistent with the participants final intervention step. Participants will also continue to complete monthly check-ins with the study coordinator to complete the Composite Asthma Severity Index, the Asthma Control Test, and a spirometry test.

ELIGIBILITY:
Inclusion Criteria:

* Patient age between 12-18 years
* Patient is diagnosed with severe-persistent or moderate-persistent asthma per NAEPP asthma guidelines
* Patient is prescribed at least one daily inhaled controller medication or a daily combination inhaled corticosteroid and long-acting beta-agonist and a beta-agonist bronchodilator
* English fluency for patient, caregiver, and clinician

Exclusion Criteria:

* Significant cognitive deficits that may interfere with comprehension per medical team or chart review.
* Diagnosis of serious mental illness (e.g., schizophrenia)
* Diagnosis of pervasive developmental disorder
* Active chronic disease apart from asthma or allergic disease (e.g. Bronchiectasis)
* Patient receives school administered daily controller medication at the time of the enrollment visit

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2018-12-07 (Actual); Primary Completion 2021-04-20 (Actual); Study Completion 2021-04-20 (Actual)

PRIMARY OUTCOMES:
Electronic Monitoring | 12 months
  The Propeller Health monitoring system includes a Bluetooth enabled sensor that attaches to the patient's inhaler. This sensor records every dose, or "puff", the patient takes and sends it to a corresponding online database that is accessible to study staff. Participants will be given this sensor at baseline.

SECONDARY OUTCOMES:
Lung Function Assessment | Baseline assessment and then once a month for 12 months
  The mobile spirometer records multiple parameters of the patient's lung function including forced expiratory volume, peak expiratory flow, forced vital capacity, and forced expiratory flow. The spirometer sends the values to the corresponding mobile phone application, Propeller Health, which is directly accessible to the patient.
Composite Asthma Severity Index (CASI) | Baseline assessment and then once a month for 12 months
  The participants' composite asthma severity index score will be calculated through the TreatSmart program. TreatSmart will be used to determine the participant's symptom burden, health care utilization, systemic corticosteroid use, and current medication use to determine the level of asthma severity/control the participant has. The program also makes an initial treatment recommendation based on the National Asthma Education and Prevention Program (NAEPP asthma guidelines). Individuals are placed in Step 1 through Step 6 depending on the strength and frequency of their inhaled corticosteroid (1 being low dose and 6 being a high dose). In addition, individuals are categorized as very poorly controlled, not well controlled, or well controlled based on how frequently they have had asthma symptoms or used their rescue inhaler, gone to the hospital or urgent care, or received steroids for asthma symptoms.
Asthma Control Test (ACT) | Baseline assessment and then once a month for 12 months
  The ACT will be used as a measure of disease severity in this study. The ACT is a 5-question scoring tool designed for patients with asthma who are 12 years and older. The questions ask the patient to rate their asthma severity, symptom frequency, control, and inhaler use on a scale of 1-5. The total score is calculated by the sum of each response, which determines how well-controlled the patient's asthma is on a scale from 5-25.
Attendance/Participation rates | 12 months
  Participation rates will be measured 3 different ways. The first measure will be how often participants accessed the electronic material (educational materials and/or Propeller Health app), the second measure will be how many responses to directive text messaging were received, and the third measure will be attendance to the telehealth sessions.
Feasibility/Acceptability Questionnaire | 5 months
  A 5-31 item measure of format, content, length, skills and acceptability of the intervention will be given to participants in the form of a questionnaire at the end of each step and the end of the study. The feasibility section is on a scale of 0 to 4, 0 being the worst and 4 being the best. The acceptability questionnaire is on a scale from 'Not at all' to 'Very,' 'Not at all' being the worst and 'Very' being the best.
System Usability Scale | 5 months
  A 10 item, Likert scale giving a global view of usability will be given to participants in the form of a questionnaire at the end of each step and at the end of the study. The scale ranges from 'Strongly Disagree' to 'Strongly Agree, with half of the items reverse scored.
Acceptability of Intervention Measure (AIM) | At 5 months
  A 4 item measure of participants' belief that the intervention is acceptable will be given at the end of the study. Participants respond to each statement on a 5 point Likert scale (1= Completely Disagree, 5= Completely Agree).
Intervention Appropriateness Measure (IAM) | At 5 months
  A 4 item measure of participants' perception that the intervention is appropriate will be given at the end of the study. Participants respond to each statement on a 5 point Likert scale (1= Completely Disagree, 5= Completely Agree).
Feasibility of Intervention Measure (FIM) | At 5 months
  A 4 item measure of participants' belief that the intervention is feasible will be given at the end of the study. Participants respond to each statement on a 5 point Likert scale (1= Completely Disagree, 5= Completely Agree).
Treatment Fidelity | 12 months
  Treatment fidelity needed for the intervention will be assessed. Treatment fidelity will be assessed through fidelity checklists created specifically for each intervention session.
Time Needed for Intervention | 12 months
  Sessions will be timed and the number of weeks to complete the session will be tracked to determine the average length of time needed for the intervention.
Perceived Characteristics of Intervention Scale | At 12 months
  19 item measure of interventionist views toward the study intervention.

OTHER OUTCOMES:
Behavior Assessment System for Children-Third Edition, Self-report of Personality (BASC-3-SRP-A | Baseline assessment and at 5 months
  The BASC-3 is a widely used, reliable (α= 0.94 - 0.96 , test-retest r= 0.81 -0.82), and valid inventory to assess emotional and behavioral symptoms in adolescents and young adults (ages 13-21).
Adolescent Barriers to Medication Scales (AMBS) | Baseline Assessment
  The AMBS is an 18-item validated measure of perceived barriers to medication adherence in adolescents.
Technology-based Experience of Need Satisfaction- Interface questionnaire (TENS-Interface) | Baseline assessment and then at 2 months
  A 15- item measure of participant's competence, autonomy, and relatedness in using technology. Participants rate their level of agreement to each statement on a 5- point Likert scale (1= Do Not Agree, 5= Strongly Agree).
Autonomy and Competence in Technology Adoption Questionnaire (ACTA) | Baseline Assessment
  A 10-item measure of why people adopt use of a technology (i.e. download an app, register with a website, purchase a wearable device, etc.).Participants respond to self-regulation statements on a scale of 1 to 5, 1 being 'not at all true' and 5 being 'very true.'
Technology-based Experience of Need Satisfaction- Task questionnaire (TENS- Task) | Baseline assessment and then at 2 months
  An 8-item measure of participant's competence, autonomy, and relatedness in managing their asthma using technology. Participants rate their level of agreement to each statement on a 5- point Likert scale (1= Do Not Agree, 5= Strongly Agree).
Technology Effects on Need Satisfaction in Life (TENS- Life) | Baseline assessment and then at 2 months
  The TENS-Life is a 10- item measure of the extent to which a user perceives that the use of a particular technology has had an influence on the satisfaction of basic psychological needs in their life. Participants rate their level of agreement to each statement on a 5- point Likert scale (1= Do Not Agree, 5= Strongly Agree).
Knowledge Questionnaire | Baseline Assessment
  A 13-item questionnaire assessing individual's knowledge of asthma symptoms, triggers, and medications. Participants rate their level of agreement to each statement on a scale from 'Strongly Agree' to 'Strongly Disagree.' This questionnaire will be completed at the baseline visit.
Hardship Questionnaire | Baseline Assessment
  A 19-item validated questionnaire assessing the financial strain of individuals within a household.

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Medical Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided